CLINICAL TRIAL: NCT04086953
Title: Validation of a Walk-Time Limit Test (WTLT) Derived from the 6-Minute Walk Test (6-MWT) in Patients with Chronic Cardiovascular or Respiratory Diseases
Acronym: TTLM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion difficulties (44/100 patients) despite a 24-month extension. The population often presents with 2 concomitant diseases.
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC19.0134 TTLM
Record Dates: First submitted 2019-08-29; First posted 2019-09-12 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Cardiovascular Insufficiency
Keywords: Exercise Test; Walking Test; Chronic Disease; Endurance Time; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Chronic Disease | interventions — Walk Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chronic Respiratory Disease Group (Experimental): Each patient receive the same intervention : 4 visits with different exercise tests.
  Visit 1: Inclusion Visit, Functional Assessment and TTLM Speed Determination (6-minute walk test x2, cardiopulmonary exercise testing on ergocycle, questionnaires and accelerometer)
  Visit 2 : Functional Evaluation and Shuttle Tests (ISWT, ESWT, Speed tests on 4m, Quadriceps muscle strength)
  Visit 3 : Feasibility of the WTLT (WTLT x2 or 3)
  Visit 4 : Reproducibility of the WTLT (WTLT x2) Specific measures for COPD subjects : Respiratory Functional Assessment and Dyspnea questionnaire
  Interventions: Diagnostic Test: 6-minute walk test; Diagnostic Test: Walk-Time Limit Tes; Diagnostic Test: Incremental shuttle walk test; Diagnostic Test: Endurance shuttle walk test; Diagnostic Test: Respiratory Functional Assessment
- Cardiovascular diseases Group (Experimental): Each patient receive the same intervention : 4 visits with different tests.
  Visit 1: Inclusion Visit, Functional Assessment and TTLM Speed Determination (6-minute walk test x2, cardiopulmonary exercise testing on ergocycle,, questionnaires and accelerometer)
  Visit 2 : Functional Evaluation and Shuttle Tests (ISWT, ESWT, Speed tests on 4m, Quadriceps muscle strength)
  Visit 3 : Feasibility of the WTLT (WTLT x2 or 3)
  Visit 4 : Reproducibility of the WTLT (WTLT x2)
  Interventions: Diagnostic Test: 6-minute walk test; Diagnostic Test: Walk-Time Limit Tes; Diagnostic Test: Incremental shuttle walk test; Diagnostic Test: Endurance shuttle walk test

INTERVENTIONS:
Diagnostic Test: 6-minute walk test — This test is carried out in a 30-meter long walking corridor with two cones placed at the ends of the course and representing the turning zones
Diagnostic Test: Walk-Time Limit Tes — Endurance test where the patient must walk at the same speed during the whole test (time limit). The test is carried out in a corridor 10 meter long.
Diagnostic Test: Incremental shuttle walk test — Incremental walking test suitable for patients with chronic respiratory diseases. To perform this test, it is necessary to have a 10-meter walking corridor. The walking speed is dictated by a sound signal previously recorded. Every minute, the time between each beep is decreased and therefore the walking speed increased. The increment is 0.17m / sec every minute. Shifting to a higher speed is indicated by a triple beep. At most, the ISWT includes 12 speed levels.
Diagnostic Test: Endurance shuttle walk test — Constant load endurance running test performed on the same 10 meter run as the ISWT.
  The patient is walking at a constant speed imposed by the audio beeps as for the ISWT. The objective of this test is to maintain the imposed walking speed as long as possible. The speed is calculated from the ISWT.
Diagnostic Test: Respiratory Functional Assessment — Forced vital capacity, total lung capacity, forced expiratory volume measured during the first second of forced expiration, and carbon monoxide diffusion capacity will be measured by plethysmographic examination and spirometry.
  Arms: Chronic Respiratory Disease Group

SUMMARY:
Many exercise tests are commonly used to evaluate the changes of exercise tolerance following rehabilitation programs in patients with chronic respiratory diseases.

Among the tests (6-MWT, incremental test, ...), the literature seems to indicate that endurance time is the most responsive parameter for detecting and quantifying changes in exercise capacity following a rehabilitation program. Although its clinical interest is undeniable, the endurance shuttle walking test is rarely used because it requires the prior performance of two incremental shuttle walking tests to determine the walking speed imposed on the patient.

In this protocol, we propose to test a Walk-Time Limit Test (WTLT) derived from the 6-minute walk test (6-MWT) and based on the average walking speed achieved in this test commonly used in the follow-up of patients with chronic diseases.

TTLM validation would improve the functional assessment of patients with chronic diseases while limiting the number of exercise tests.

DETAILED DESCRIPTION:
Each patient will perform 4 visits over a period of 4-week. Fifty subjects with COPD and fifty subjects with heart failure will be recruited for the same protocol.

During the first visit, the subject will realize two 6-MWT and a cardiopulmonary exercise test on ergocycle with the measure of cardiorespiratory parameters. We will evaluate the physical activity during daily life using an accelerometer and we will use several questionnaires to measure the quality of life, the motivation to physical activities and symptoms.

During the second visit, the subject will realize a 4-meter walk test, two incremental shuttle walk tests (ISWT), an endurance shuttle walk test (ESWT) and a test with dynamometer to measure the quadriceps strength.

During the third and fourth visits, the subject realize two or three endurance walking tests (Walk-Time Limit Test - WTLT) at a walking speed equivalent to the mean speed realize during the better 6MWT (visit 1)

ELIGIBILITY:
Inclusion Criteria:

* Chronic Respiratory Disease Group:

  * Diagnosis of COPD with FEV1 corresponding to stages GOLD II or III (50-80% predicted or 30-50% predicted, respectively).
  * Patient's agreement
  * Being older than 18
  * Stable treatment for 3 months
  * Subjects affiliated with social security
* Group cardiovascular diseases:

  * Diagnosis of heart failure or stable coronary artery disease with NYHA Class II stage.
  * Patient's agreement
  * Being older than 18
  * Stable treatment for 3 months
  * Subjects affiliated with social security

Exclusion Criteria:

* Any medical contraindications to the practice of a suitable physical activity
* Presence of muscle, joint and / or neurological comorbidities affecting motor skills and test performance.
* Refusal of the patient
* Subject under guardianship or curatorship
* Subject aged over 80 at the time of inclusion
* Realization of a rehabilitation program during the study period
* Subject under resting oxygen therapy
* Diagnosis of heart failure, coronary artery disease or any cardiovascular pathology that required surgery.
* Diagnosis of an associated chronic respiratory disease, such as asthma, pulmonary arterial hypertension or interstitial lung disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Endurance time | 4 weeks
  The patient walks at the same speed during the entire test in a corridor 10 meters long around studs placed at a distance of 9m

SECONDARY OUTCOMES:
Maximum speed measured at the ISWT | 0 day
  Realization of ISWT (Incremental shuttle walk test) : The walking speed is dictated by a sound signal previously recorded. Every minute, the time between each beep is decreased and therefore the walking speed increased. The increment is 0.17m / sec every minute. At the maximum, the ISWT has 12 speed levels ranging from 1.8 km/h (start of test) to approximately 8.5 km/h
Walking distance to 6-MWT | 0 day
  Realization of 6-MWT
Number of steps by day (accelerometer) | 7 days
  wearing an accelerometer
Maximum speed measured (4-meter walk test) | 0 day
  Realization of 4-meter walk test
Oxygen consumption | 1 day
  VO2 ( in L/min)
Dyspnea and leg fatigue during tests after WTLT | 7 days
  Assessment thanks to a score between 0 and 10 given by the patient before and after WTLT
Forced expiratory volume per second | 0 Day
  FEVS (in L)
Quadriceps strength | 0 day
  Manual dynamometer
Score of motivation thanks to Behavourial Regulation and Exercise Questionnaire 2 (BREQ-2) | 0 day
  The answer to questions goes from 0 to 4 with 0 (not at all), 2 (sometimes it's true) and 4 (yes, absolutely).
Following of the quality of life | 0 day
  The Short Form 36 (SF36) is used to evaluate the quality of life. The SF36 scale includes 36 items divided into 8 dimensions (physical functioning, role limitations related to physical health, physical pain, general health, vitality [energy / fatigue].
carbon dioxide production | 1 day
  VCO2 ( in L/min)
breathing frequency | 1 day
  RF (in breaths/min)
heart rate | 1 day
  BPM (in beat per minute)
Forced Vital Capacity | 0 day
  FVC (in L)
Diffusing capacity for carbon monoxide | 0 day
  DLCO (in mL/min/mmHg)
Total Lung Capacity | 0 day
  TLC (in L)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Brest, Brest, France, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.